CLINICAL TRIAL: NCT06563479
Title: Phase III Randomized and Double-blinded Trial of De-escalated Radiation in FMISO PET-selected Good Risk Versus Standard of Care Radiation in Unselected HPV Positive Oropharyngeal Cancer
Brief Title: A Study Comparing Personalized Radiation Therapy With Standard Radiation Therapy in People With HPV-Positive Throat Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-200
Record Dates: First submitted 2024-08-19; First posted 2024-08-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: HPV-Related Squamous Cell Carcinoma
Keywords: oropharynx; tonsil; base of the tongue; oropharyngeal walls; radiation treatments; cisplatin; 24-200
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Personalized Chemoradiation Therapy (Experimental): Patient without evidence of hypoxia will receive 30Gy in 2Gy per fraction. Concurrent chemotherapy will be given as per guidelines. After completion of chemotherapy and radiation therapy, a 4 month (+/- 4 weeks) posttreatment standard FDG PET/CT scan will be performed and if there is persistent disease, standard neck dissection will be performed. Further standard of care will be given pending pathologic findings.1. Hypoxia negative: The entire target volume which includes GTV and CTV will receive 30Gy in 2 Gy per fraction over 15 days (PTV30). 2. Hypoxia positive (same as the standard of care): The CTV will receive 50Gy in 2Gy per fraction over 25 days. This is name PTV50 and will receive 50Gy in 2Gy per fraction over 25 days. The GTV will receive an additional boost of 20Gy in 2 Gy per fraction so that the total PTV70 dose is 70Gy.
  Interventions: Diagnostic Test: FMISO-PET Scan; Combination Product: Chemoradiation; Other: Assessments
- Standard Chemoradiation Therapy (Active Comparator): Patient will receive 70Gy in 2Gy per fraction regardless of hypoxia status. Concurrent chemotherapy will be given as per guidelines. After completion of chemotherapy and radiation therapy, a 4 month (+/- 4 weeks) posttreatment standard FDG PET/CT scan will be performed and if there is persistent disease, standard neck dissection will be performed. Further standard of care will be given pending pathologic findings.
  Interventions: Diagnostic Test: FMISO-PET Scan; Combination Product: Chemoradiation; Other: Assessments

INTERVENTIONS:
Diagnostic Test: FMISO-PET Scan — Patients will undergo 18F-FMISO scan (only 1 injection) that occurs at week two of radiation treatment, typically day 10 but a window of 8-10 radiation treatment days* after start of radiation is allowed.
Combination Product: Chemoradiation — 30 Gy or 70 Gy of radiation in combination with standard chemotherapy (cisplatin, carboplatin, and 5-FU)
  Arms: Personalized Chemoradiation Therapy
Combination Product: Chemoradiation — 70 Gy of radiation in combination with standard chemotherapy (cisplatin, carboplatin, and 5-FU)
  Arms: Standard Chemoradiation Therapy
Other: Assessments — EQ-5D-5L (5 questions); 2. MDADI-HN (total of 20 questions); 3. COST-FACIT (total of 12 questions).

SUMMARY:
The researchers are doing this study to find out if a personalized approach to chemoradiation therapy (which may include a lower dose of radiation) is as effective as the standard chemoradiation therapy in people with HPV-positive throat cancer. Other purposes of this study include looking at the following:

* Whether a lower dose of radiation in combination with standard chemotherapy causes fewer side effects than the standard dose of radiation therapy in combination with standard chemotherapy
* How the study approaches (lower dose of radiation therapy + standard chemotherapy and standard dose of radiation therapy + standard chemotherapy) affect participants' quality of life. The researchers will measure quality of life by having participants fill out questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of HPV associated squamous cell carcinoma of the oropharynx (tonsil, base of tongue, or oropharyngeal walls) or squamous cell carcinoma with an unknown primary. Surgical removal of primary site is allowed.
* Patients must test positive for both p16 expression (70% nuclear and cytoplasm expression; Ventana Medical Systems) and mRNA HPV in situ hybridization (RNAscope® 2.5 HD Reagent kit (Advanced Cell Diagnostics, Inc, Hayward, CA). Any CLIA certified testing method can be used.
* Clinical stage Tx-2, N1-2c (AJCC, 7th ed.) without evidence of distant metastasis based on FDG PET/CT.
* ECOG Performance Status of 0-1 or KPS >/=70
* Age ≥ 18
* Adequate hematologic function within 30 days prior to registration, defined as follows:

  * White Blood Count (WBC) ≥ 2 K/mcL
  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3
  * Platelets ≥ 100,000 cells/mm^3
  * Hemoglobin ≥ 10.0 g/dl
* Adequate renal function within 30 days prior to registration, defined as follows:

  o Serum creatinine < 1.5 mg/dl or creatinine clearance (CC) ≥ 50 ml/min determined by 24-hour collection or estimated by Cockcroft-Gault formula: CCr male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)] CCr female = 0.85 x (CrCl male)
* Negative serum pregnancy test within 14 days prior to registration for women of childbearing potential
* The patient must provide study-specific informed consent prior to study entry
* Optional section of the protocol: Patients must be able to undergo MRI scans, i.e. not claustrophobic

Exclusion Criteria:

* Patients with prior head and neck radiation therapy where there is >30% overlap with the current head and neck radiation fields. Exceptions can be made if determined by the PI/Co-PI that the patient can proceed with protocol activities
* Patients whose tumors are borderline T4 based on anterior tumor extension to the extrinsic muscles of the tongue
* Patients with simultaneous primary cancers outside of the oropharynx

  o Note: Exceptions can be made for patients with simultaneous primaries outside the oropharynx if determined by the PI/Co-PI the patient can proceed with protocol activities
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for 3 years or if cure rate from treatment at 5 years to be 90% or greater

  o Note: Exceptions can be made for patients with prior malignancies outside the oropharynx if determined by the PI/Co-PI the patient can proceed with protocol activities.
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* No particle therapy
* Patients who are deemed non-compliant to all the protocol related activities
* Contraindications to receive either cisplatin or the combination of carboplatin/5-fluorouracil at the prescribed doses.
* Severe, active co-morbidity defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration
  * Hepatic Insufficiency resulting in clinical jaundice and/or coagulation defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2 years
  The measurement of survival will be evaluated as a time from randomization to events endpoint (i.e., death due to any cause) so that censored data are allowed. To assess the overall survival rate, Kaplan-Meier estimates will be calculated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Hartford Healthcare (Data Collection Only), Hartford, Connecticut
  - Baptist Alliance MCI (Data Collection Only), Miami, Florida
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm